CLINICAL TRIAL: NCT04168411
Title: A Prospective Comparison of Clinical, Functional, and Isokinetic Outcomes Between Short Leg Cast Immobilization and Symptomatic Treatment in Tuberosity Fractures of the Proximal Fifth Metatarsal
Brief Title: Comparison Different Method Treatment in Tuberosity Fractures of the Proximal Fifth Metatarsal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Serkan Bayram, Medical Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/536
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Muscle Weakness; Metatarsal Fracture; Healing Fracture of Bone
Keywords: metatarsal, fracture, muscle weakness, isokinetic test,
MeSH Terms: conditions — Muscle Weakness; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic treatment group (Experimental): The patients were allocated to wear a double layered elasticated bandage for treatment 5th metatarsal base fractures (Zone 1).
  Interventions: Procedure: Symptomatic Treatment
- Cast group (Active Comparator): The patients were given a below-knee cast for treatment 5th metatarsal base fractures (Zone 1).
  Interventions: Procedure: Symptomatic Treatment

INTERVENTIONS:
Procedure: Symptomatic Treatment — Conservative treatment methods of tuberosity fractures of the proximal fifth metatarsal

SUMMARY:
Fracture of the base of the fifth metatarsal is one of the most common injuries in ankle trauma. There are many conservative treatment protocols for fifth metatarsal base fractures which have up to 99% success. Short leg cast and walking boot are conservative treatment methods that aim to prevent weight-bearing. There are many different conservative treatment methods that allow weight-bearing such as an elastic bandage. There was no significant difference between cast and symptomatic treatment in the previous studies. Muscle atrophy developing after immobilization with cast may adversely affect the daily activities of the patient in the first few months. However, there was no study comparing the effect of these two treatment methods on ankle muscle strength.

In this study, the investigators compared the strength of the ınjured and healthy ankle muscle when symptomatic and cast treatment methods are applied to patients with tuberosity fractures of proximal fifty metatars. In addition, patients' functional, clinic and radiological outcomes were also compared.

DETAILED DESCRIPTION:
We prospectively treated 73 patients with 5th metatarsal base fractures (Zone 1) who came to the emergency department. Patients were allocated to a treatment group using an electronic random number generator. The generation of an even number randomized the participant to a below-knee cast, and an odd number to a double-layered elasticated bandage. In all, patients were allocated to wear a double layered elasticated bandage (group 1) applied by S.B and patients were given a below-knee cast (group 2) applied by D.K. Duration of both treatments were for four weeks and the cast removed in that time in our clinic. This reference form of treatment was the same as in previous reports.

The non-injured extremity was measured with isokinetic test at initial injury time for evaluation of side effect of immobilization after treatment. At that time, patients were asked for height, weight and pain scores. Body muscle index was calculated for all patients. Tobacco using was also asked.To measure clinical outcomes, using the validated Visual Analogue Scale Foot and Ankle (VAS-FA) score [7] and The EuroQol-5D visual analogue scale (EQ-5D VAS) score were used [8]. The VAS-FA score ranges from 0 to 100 points: higher scores indicate a better functional outcome. EQ-5D VAS score was used as a secondary outcome measure: this ranges from 0 to 100. Baseline functional scores were collected at the time of consult in the clinic.

Both ankle plantar-dorsiflexors and inversion-eversion'strength (peak torque %BW (Body Weight)) were measured with an isokinetic dynamometer (Cybex Humac Norm, CA, USA) at Isokinetic Test Laboratory of Sports Medicine in the Istanbul Medical Faculty. Test procedure was performed by the same investigator (T.Ş) in all cases for ensuring standardization. The muscle strength can be defined as the capacity of a muscle to withstand great force.

Injured extremity values were compared with non-injured extremity. The non-injured extremity was measured at initial injury time for evaluation of side effect of both treatment methods. The tests were started with non-injured sides of the patients and measurements at low angular velocity. The dynamometer was calibrated at the beginning of each testing session. Subjects were tested in prone position and stabilized in the exercise chair as per the manufacturer's recommendation. The anatomical axis of the ankle was aligned with the axis of the dynamometer while the foot was secured to the foot plate with velcros. Proximal stabilization was achieved with the straps at the thigh and calf. In the test, dorsiflexion-plantarflexion and inversion-eversion peak torque force (strength) measurements were performed in 3 trials and 3 tests repetitions at 30 degrees/sec angular speed for both side of the patient.

All of the patients were given follow-up appointments at 2, 4, 8, 12 and 24 week interval at our clinic. Radiographs were similarly scheduled for 4, 8, and 12 week intervals to assess bony healing. However, functional outcomes and isokinetic test was applied also at 24 week control. At second visit, isokinetic test was not applied. These studies were started on fixed ground and then continued on moving boards. Standard rehabilitation program was given for all patients each group included joint mobilizations, passive stretching, electrotherapy-ice compression for pain relieving and ankle proprioceptive exercises, as considered necessary by same author (T.Ş).

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Acute (presented within one week of injury) Zone 1 fractures of fifth metatarsi

Exclusion Criteria:

* Zone 2-3 fractures
* Diabetes mellitus
* Osteoporotic bone (T score<-2.5),
* History of osteoporotic drug therapy,
* Other lower extremity any fracture,
* Previous foot surgery or fracture in both lower extremity,
* Chronic fracture, pathological fracture,
* Aged over 65 years (congruity of muscle strength test)
* Open fracture

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Changed of Baseline Isokinetic Muscle Strength at 6 months | Isokinetic Muscle Strength test was scheduled for baseline, 4, 8,12 and 24 week intervals to assess ankle muscle strength
  Both ankle plantar-dorsiflexion muscle strength and inversion-eversion muscle strength (peak torque %BW (Body Weight)) were measured with an isokinetic dynamometer (Cybex Humac Norm, CA, USA) at Isokinetic Test Laboratory of Sports Medicine in the Istanbul Medical Faculty. Test procedure was performed by the same investigator in all cases for ensuring standardization. The muscle strength can be defined as the capacity of a muscle to withstand great force. Injured extremity values were compared with healthy extremity. he healthy extremity was measured at initial injury time for evaluation of side effect of both treatment methods.

SECONDARY OUTCOMES:
Changed of Baseline VAS-FA Scores at 6 months | baseline, 2, 4, 8,12 and 24 weeks follow-up visit
  The investigators was measured clinical outcomes, using the validated "Visual Analogue Scale Foot and Ankle (VAS-FA) Score". VAS-FA score is numbered from 0 to 100. 100 is the best health and 0 is the worst health.
Changed of Baseline EuroQol-5D VAS Scores at 6 months | baseline, 2nd, 4th, 8th,12th and 24th week follow-up visit
  The investigators was measured clinical outcomes using The EuroQol-5D visual analogue scale (EQ-5D VAS). (EQ-5D VAS is numbered from 0 to 100. 100 is the best health and 0 is the worst health.

OTHER OUTCOMES:
Number of Days with using an assistive device | through study completion, an average of 6 months
  Patients use the Canadian sticks while walking for decrease their pain level. The time of the using assistive device was investigated and compared between both groups.
Number of Days with a take of analgesia | through study completion, an average of 6 months
  Patients take the pills for their pain. Our drug choose is paracetamol for patients. The time of take of drug was investigated and compared between both groups.
Number of Days with unable to work | through study completion, an average of 6 months
  The time taken of unable to work was investigated and compared between both groups.
Rates of Complications | through study completion, an average of 6 months
  Every treatment method has got a lot of complications. The complications of both treatment methods were investigated and noted. The complication rates of the treatment methods were compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Akgul, MD, Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)